CLINICAL TRIAL: NCT06851689
Title: Correlation Between Shoulder Rotation Torque and Hand Grip Strength in University Teaching Staff
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abanoub Emeil Melad Sedarous Michael, principle investigator, Cairo University
Other Study IDs: P.T.REC/012/005456
Record Dates: First submitted 2025-02-23; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hand Grip Strength; Torque
Keywords: hand grip; shoulder torque; academic staff

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Jamar handheld dynamometer — Jamar handheld dynamometer to asses hand grip strength
Device: Biodex isokinetics — Biodex isokinetics to asses torque

SUMMARY:
The aim is to reduce the incidence of hand grip weakness and shoulder rotation torque decline. this proposed study aims to suggest solutions to prevent occurring injuries

DETAILED DESCRIPTION:
Teaching is becoming a high-risk job for injuries. In recent years, there has been a growing concern about work-related musculoskeletal disorders (WMSDs) among teachers. These disorders include injuries and pain in muscles, tendons, and nerves. Studies show that teachers are more likely to experience WMSDs than people in other professions, with rates reported to be between 39% and 95%. This is a serious issue that deserves attention after being ignored for a long time.

Potential for Injury Prevention: Physical therapy and occupational health professionals can utilize this correlation to design preventive strategies. For instance, if a significant correlation exists, interventions aimed at improving shoulder torque through specific exercises could also enhance hand grip strength, thereby reducing the risk of musculoskeletal injuries among university teaching staff . Educational and Workplace Ergonomics: Insights from this correlation can inform educational institutions and workplaces about ergonomics and physical fitness programs. Implementing ergonomic practices and wellness programs that target upper body strength could potentially improve overall health outcomes and productivity among university teaching staff . One of the primary issues among university teaching staff is the prevalence of shoulder and upper limb problems. Treatment typically focuses solely on the shoulder and neglects the wrist. Workers in overhead workplaces are in a hazardous position . Ergonomic solutions should be developed to prevent muscle fatigue and decreased grip force.

The aim is to reduce the incidence of hand grip weakness and shoulder rotation torque decline.Given the fact that many injuries are preventable, this proposed study aims to suggest solutions to prevent occurring injuries. Based on the findings, recommendations could potentially decrease shoulder and hand problems and enhance the quality of life for the university teaching staff. Insufficient research has been conducted on the association between hand grip strength and shoulder muscle torque in teaching staff. Therefore, this study aims to pave the way for future research to address this critical issue. There is a gap in the literature about hand grip strength and shoulder rotation torque between university teaching staff so This study will be conducted to investigate the correlation between rotation shoulder torque and hand grip strength between university teaching staff.

ELIGIBILITY:
Inclusion Criteria:

1. University teaching staff who work full time at Misr University for Science and Technology. (average 7 hours per day)
2. Both male and female participants between 25 and 45 years of age
3. Participants without any pain or musculoskeletal disorder
4. Participants who perform overhead activities during teaching
5. The range of BMI is between 18.5-25 in the normal range
6. Both right and left handed subjects are included

Exclusion Criteria:

* 1.Recent history of shoulder, upper limb, neck or thoracic fracture or surgery

  2. Neurological disorders affecting the upper limb

  3. Regional tumor or metastasis of the upper limb

  4. Academicians with trauma or injury within the past 6 months, or known pregnancy

  5. Engagement of any vigorous exercise or work after university hours

  6.History of surgery within the past six months, epilepsy, or chronic neurologic disease

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult academic staff
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
hand grip strength | 2 months
  assess hand grip
shoulder torque | 2 months
  assess peak shoulder torque of rotator muscle

CONTACTS AND LOCATIONS:
Overall Officials: Abanoub Emeil Melad, Bachelor, Principal Investigator — Misr University for Science and Technology; Neveen Abdel-Latif, professor, Study Chair — Cairo University; Rania Reda, Ass.prof, Study Director — Cairo University; Mohamed Farouk, lecturer, Study Chair — Misr University for Science and Technology

IPD SHARING:
Plan to Share IPD: No